CLINICAL TRIAL: NCT05566405
Title: Comparative Study of the Effects of Combined Spinal Anaesthesia and General Anaesthesia on the Safety and Effectiveness of Radical Retropubic Prostatectomy in Patients With Localised Prostate Cancer
Brief Title: The Effects of Method of Anaesthesia on the Safety and Effectiveness of Radical Retropubic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sismanoglio General Hospital (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Pikramenos, Principal Investigator, Urology Resident, MD, Sismanoglio General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PN 20511/14.10.2020
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Anesthesia, General; Injections, Epidural; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anaesthesia (Active Comparator): Patients undergoing open retropubic radical prostatectomy under general anaesthesia
  Interventions: Procedure: General Anaesthesia; Procedure: Open Retropubic Radical Prostatectomy
- Combined (Epidural and Spinal) Anaesthesia (Active Comparator): Patients undergoing open retropubic radical prostatectomy under combined (epidural and spinal) anaesthesia
  Interventions: Procedure: Combined (Epidural and Spinal) Anaesthesia; Procedure: Open Retropubic Radical Prostatectomy

INTERVENTIONS:
Procedure: General Anaesthesia — All patients in the general anaesthesia group will be premedicated with intravenously administered (iv) midazolam (2mg) and fentanyl (100 mcg). Induction will be performed using intravenous propofol (2.5-3mg/kg) and lidocaine (40mg); dexamethasone 8mg, metoclopramide 10mg and omeprazole 40mg will also be administered. After successful tracheal intubation, total intravenous anaesthesia will be maintained by administering propofol (0.05 mg/kg/sec iv) and remifentanil (0.2 mcg/kg/sec iv). Pain management will be achieved by paracetamol (1g iv) and tramadol (100mg iv) whereas muscle relaxation by vecuronium (0.6 mg/kg iv).
  Arms: General Anaesthesia
Procedure: Combined (Epidural and Spinal) Anaesthesia — Combined (epidural and spinal) anaesthesia will be performed using an epidural 18G needle and a spinal 27G needle, in the L2-L3 or L3-L4 interspace. Induction will be carried out by spinal intrathecal administration of levobupivacaine (2.6-3ml of 0.5%) and mild sedation by midazolam (5mg iv in bolus). All patients will be administered dexamethasone 8mg, metoclopramide 10mg and omeprazole 40mg iv. Maintenance will be performed 75 minutes after induction and obtained using an epidural administration of levobupivacaine (4-5ml of 0.5%).
  Arms: Combined (Epidural and Spinal) Anaesthesia
Procedure: Open Retropubic Radical Prostatectomy — All patients will undergo a nerve-sparing open retropubic radical prostatectomy

SUMMARY:
Prostate cancer is one of the most commonly diagnosed neoplasm in men worldwide. The gold standard of therapy is radical prostatectomy, a wide surgical excision of the neoplasm and can be performed either open, laparoscopic or robotic. The open retropubic approach, still performed today, can be completed under either general anaesthesia or combined (spinal/epidural) anaesthesia without any clear guideline on which one should be preferred.

In this study the investigators aim to evaluate general anaesthesia and combined (spinal/ epidural) anaesthesia in patients undergoing open retropubic radical prostatectomy and define whether these may have an impact on the oncological outcome and safety of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with localised prostate cancer
* Eligible for open retropubic radical prostatectomy

Exclusion Criteria:

* Metastatic prostate cancer
* History of severe heart disease
* History of haemostasis disorders
* History of previous pelvic surgery
* History of lung disease

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Change | Peri-operatively
  Measurement of patients systolic and diastolic blood pressure during the operation and post-operatively for 72 hours.
Heart Rate Change | Peri-operatively
  Measurement of patients Heart Rate during the operation and post-operatively for 72 hours.
Surgical APGAR Score | Peri-operatively
  Calculation of the Surgical APGAR score for each patient during surgery. The lower the score, on a scale of 1-10, the worst the prognosis of the patient.
  SAS is calculated using three variables:
  * Estimated blood loss (on a 0-3 scale, 0 points >1000 ml, 1 point 601-1000ml, 2 points 101-600 ml, 3 points <100ml)
  * Lowest mean arterial pressure (on a 0-3 scale, 0 points <40 mmHg, 1 point 40-54 mmHg, 2 points 55-69 mmHg, 3 points >70 mmHg)
  * Lowest heart rate (on a 0-4 scale, 0 points >85 bpm, 1 points 76-85 bpm, 2 points 66-75 bmp, 3 points 56-65 bmp, 4 points <55 bmp) during surgery.
Blood Loss During Surgery | Peri-operatively
  Measured from suction contents intra-operatively in ml
Haemoglobin Change | Peri-operatively
  Haemoglobin measurement before the operation and at 12-, 24- and 48-hours post-operatively, in g/dL
Operation Time | Peri-operatively
  Time required for:
  * Induction of anaesthesia
  * Completion of the operation
  * Post-operative time until the patient is successfully transferred to the recovery room
Pain Assessed by the VAS Scale | Peri-operatively
  Measured using a pain Visual Analogue Scale (VAS) at 6-, 24- and 48-hours after the operation.
  VAS is a self-reporting pain scale based on a 0 to 10-point system, with each point measuring 10mm on a linear line. Every patient was asked to indicate his pain levels from "No Pain" (equals 0) to "Worst Pain Imaginable" (equals 10).
Complication Rate | Peri-operatively and up to 1 year after the operation
  Complications related to the procedure:
  * Intraoperative bleeding
  * Post-operative bleeding
  * Bowel perforation
  * Cardiovascular
  * Respiratory
  Complications related to the anaesthesia technique performed:
  * Post-operative headache
  * Nausea and vomiting
  * Any signs of potential nerve damage (manifested as inability to gain leg motility)
Change From Baseline PSA Levels at 6-months | 6 months post-operative
  Measurement of Prostatic Specific Antigen (PSA) levels at 6 to establish a PSA nadir value
Change from 6-month PSA Levels at 12-months | 12 months post-operative
  Measurement of Prostatic Specific Antigen (PSA) levels at 12 post-operation to detect any biochemical recurrence

SECONDARY OUTCOMES:
Change from Baseline Erectile Function after Radical Prostatectomy | Up to 1 year after the operation
  Measured using the International Index of Erectile Function (IIEF-5) questionnaires pre-operatively and at 3-, 6- and 12-months post-surgery.
  The test is composed of 5 questions with 5 points for each question. Patients are evaluated accordingly:
  * Score 22 or more = No Erectile Disfunction
  * Score 17-21 = Mild Erectile Disfunction
  * Score 12-16 = Mild to moderate Erectile Disfunction
  * Score 8-11 = Moderate Erectile Disfunction
  * Score 7 or less = Severe Erectile Disfunction
  Results will be:
  * Analysed and compared to evaluate any potential difference of the two methods of anaesthesia, on post-operational erectile function
  * Analysed comparing pre-operation with post-operation questioners overall, to evaluate erectile disfunction after radical prostatectomy regardless of method of anaesthesia.
Post-operative Urinary Incontinence | 1 year after the operation
  Measured using the International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form at 12 months post-surgery.
  The Questionnaire is consisted of 4 questions:
  * Frequency "How often do you leak urine?" on a scale of 0 (never) to 5 (all the time)
  * Amount of leakage "How much urine do you leak?" on a scale to 0 (none) to 3 (a large amount)
  * Overall impact on quality of life "How much does it interfere with your life?" on a scale of 0 (not at all) to 10 (a great deal)
  * Timing of leakage "When does urine leak?"
Total Hospital Stay | Peri-operative
  Days until patient discharge from the hospital.
Patient Satisfaction Assessed by the Short Assessment of Patient Satisfaction (SAPS) Questionnaire | Peri-operative
  Satisfaction, using the Short Assessment of Patient Satisfaction (SAPS) Questionnaire, is measured in a scale of 0 to 28, with 0 to 10 equals to "Very Dissatisfied", 11-18 equals to "Dissatisfied", 19-26 equals to "Satisfied" and 27-28 equals to "Very Satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Pikramenos, MD, Principal Investigator — 2nd Urology Department, Sismanoglio Hospital, National and Kapodistrian University of Athens; Iraklis Mitsogiannis, Assoc. Prof., Study Director — 2nd Urology Department, Sismanoglio Hospital, National and Kapodistrian University of Athens; Ioannis Varkarakis, Prof., Study Chair — 2nd Urology Department, Sismanoglio Hospital, National and Kapodistrian University of Athens; Athanasios Papatsoris, Prof., Study Chair — 2nd Urology Department, Sismanoglio Hospital, National and Kapodistrian University of Athens
Locations (1):
- Sismanoglio General Hospital, Marousi, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: On reasonable request after completion of study and analysis.
Access Criteria: Any medical researcher on an official capacity will be eligible to submit a request to the primary investigator of the study. Requests will be considered in due time and relevant information released accordingly.

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Hatzinger M, Hubmann R, Moll F, Sohn M. [The history of prostate cancer from the beginning to DaVinci]. Aktuelle Urol. 2012 Jul;43(4):228-30. doi: 10.1055/s-0032-1324651. German. PMID 23035261
- [Background] Lepor H. A review of surgical techniques for radical prostatectomy. Rev Urol. 2005;7 Suppl 2(Suppl 2):S11-7. PMID 16985892
- [Background] Gawande AA, Kwaan MR, Regenbogen SE, Lipsitz SA, Zinner MJ. An Apgar score for surgery. J Am Coll Surg. 2007 Feb;204(2):201-8. doi: 10.1016/j.jamcollsurg.2006.11.011. Epub 2006 Dec 27. PMID 17254923
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Hinkelbein J, Lamperti M, Akeson J, Santos J, Costa J, De Robertis E, Longrois D, Novak-Jankovic V, Petrini F, Struys MMRF, Veyckemans F, Fuchs-Buder T, Fitzgerald R. European Society of Anaesthesiology and European Board of Anaesthesiology guidelines for procedural sedation and analgesia in adults. Eur J Anaesthesiol. 2018 Jan;35(1):6-24. doi: 10.1097/EJA.0000000000000683. PMID 28877145
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Hawthorne G, Sansoni J, Hayes L, Marosszeky N, Sansoni E. Measuring patient satisfaction with health care treatment using the Short Assessment of Patient Satisfaction measure delivered superior and robust satisfaction estimates. J Clin Epidemiol. 2014 May;67(5):527-37. doi: 10.1016/j.jclinepi.2013.12.010. PMID 24698296